CLINICAL TRIAL: NCT02886052
Title: Therapist Guided Internet Cognitive Behavioral Therapy (ICBT) for Insomnia for Bereaved Parents: a Randomized Controlled Trial (RCT)
Brief Title: Internet-based Cognitive Behavior Therapy for Insomnia for Parents Who Have Lost a Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Josefin Sveen, PhD, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ2015-0021
Record Dates: First submitted 2016-08-15; First posted 2016-09-01 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Insomnia; Bereavement
Keywords: Cognitive behavior therapy; Internet treatment; Self-help treatment; Insomnia; ICBT; CBT-i; Bereavement
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICBT for insomnia (Experimental): Therapist guided Internet-CBT for insomnia
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia
- Active control (Active Comparator): Written information on sleep, insomnia, and sleep hygiene
  Interventions: Other: Active control

INTERVENTIONS:
Behavioral: Therapist guided Internet-CBT for insomnia
  Arms: ICBT for insomnia
Other: Active control
  Arms: Active control

SUMMARY:
The purpose of this project is to evaluate an Internet-based Cognitive Behavioral Therapy (ICBT) for bereaved parents with insomnia. Participants are randomized to either a therapist guided ICBT or to an active control who receives written information on sleep, insomnia, and sleep hygiene. The primary purpose is to evaluate changes in insomnia severity for treatment compared control, after treatment and at 9 and 18 months follow up. A secondary purpose is to evaluate changes in symptoms of complicated grief and depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia according to DSM-5
* Enough Swedish language skills

Exclusion Criteria:

* Other sleep disorders that require other treatment (e.g. sleep apnea)
* Somatic or psychiatric conditions requiring acute care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in Insomnia Severity Index, ISI | 0, 9 and 18 months after treatment
  7-item, self-rated questionnaire measuring change in insomnia severity.

SECONDARY OUTCOMES:
Change (from baseline) in Montgomery Asberg Depression Rating Scale, MADRS-S | 0, 9 and 18 months after treatment
  The MADRS-S is a 9-item self-rated measure of change in depression severity.
Change (from baseline) in Prolonged Grief Disorder, PG-13 | 0, 9 and 18 months after treatment
  13-item, self-rated measure of prolonged grief disorder
Change (from baseline) in PTSD Checklist for DSM-5 , PCL-5 | 0, 9 and 18 months after treatment
  20-item, self-rated measure of posttraumatic stress disorder
Change (from baseline) in Generalised Anxiety Disorder Assessment, GAD-7 | 0, 9 and 18 months after treatment
  7-item, self-rated measure of anxiety symptoms
Change (from baseline) in Utrecht Grief Rumination Scale, UGRS | 0, 9 and 18 months after treatment
  15-item, self-rated measure of grief rumination

IPD SHARING:
Plan to Share IPD: No